CLINICAL TRIAL: NCT01686867
Title: Feasibility Intervention Trial of Two Types of Improved Cookstoves in Three Developing Countries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); National Institutes of Health (NIH) (NIH); Brown University (Other); Moi University (Other); Asociacion Benefica Prisma (Other); Nepal Nutrition Intervention Project Sarlahi (Other)
Responsible Party: Principal Investigator, William Checkley, Assistant Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: COCINAS; HHSN268200900033C (Other Grant/Funding Number: United States National Institutes of Health)
Record Dates: First submitted 2012-09-10; First posted 2012-09-18 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Poisoning by Carbon Monoxide From Domestic Fuels; Respiratory Conditions Due to Other External Agents
Keywords: improved cookstove; ventilated cookstove; behavior change; adoption; indoor air pollution; DLCO; spirometry; biomass fuel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Commercially-made followed by locally-made improved cookstove (Experimental): Following a four month run-in period using their traditional, open-fire cookstoves, the investigators will install a commercially-made improved, ventilated cookstove (Envirofit G-3300/G-3355) in each patient's kitchen. Four months later the investigators will install a locally-made improved, ventilated cookstove in each patient's kitchen. During each of the two periods, the investigators will request that the patient uses the improved, ventilated cookstove installed for that period.
  Interventions: Device: Improved, ventilated cookstove
- Locally-made followed by commercially-made improved cookstove (Experimental): Following a four month run-in period using their traditional, open-fire cookstoves, the investigators will install a locally-made improved, ventilated cookstove in each patient's kitchen. Four months later the investigators will install a commercially-made improved, ventilated cookstove (Envirofit G-3300/G-3355) in each patient's kitchen. During each of the two periods, the investigators will request that the patient uses the improved, ventilated cookstove installed for that period.
  Interventions: Device: Improved, ventilated cookstove

INTERVENTIONS:
Device: Improved, ventilated cookstove — An improved, ventilated cookstove incorporates the following key elements: burner openings customized to the size and shape of the cooking utensils; a flue designed to draw air into the fire box and pass it out through a chimney; a chimney, vented to the exterior, of adequate height to create a draft; an exterior port that has bidirectional openings to prevent the backflow of smoke and an access port for the chimney that permits cleaning.
  The investigators piloted cookstoves prior to the trial and compared their ability to reduce indoor air pollution, the reliability between cookstoves of the same type, the functionality over time, preferences and cultural compatibility, and cost. The investigators selected the the Envirofit G-3300/3355, a modified Stovetec cookstove with a chimney and a locally-made improved, ventilated cookstove for use in the trial.

SUMMARY:
The underlying concept behind this feasibility trial is to achieve a reduction in indoor smoke from biomass fuels and minimize changes in cooking practices such that it prompts one of the two improved, ventilated cookstoves to be the selection of choice. Typical fuel sources used in developing countries include wood, dried dung, and agricultural waste. The investigators propose to reduce indoor air pollution by replacing the household traditional cookstove with an improved design that incorporates the following key elements:

* Burner openings customized to the size and shape of the cooking vessels in the home.
* Flue designed to draw air into the fire box under the cooking pots and pass it out through a chimney.
* A chimney with adequate height to create a draft and vented to the exterior.
* An exterior port that has bidirectional openings to prevent backflow of smoke.
* An access port for the chimney that permits cleaning of soot.

The investigators propose to use two types of improved cookstoves that meet these criteria. As part of piloting activities, the investigators will test several different types of commercially-available cookstoves with a chimney, and we may also want to test a locally-made improved cookstove. The investigators want to evaluate those designs by comparing their ability to reduce indoor air pollution, the reliability between cookstoves of the same type, the functioning over time, the logistics of import/build locally, preferences and cultural compatibility, and costs. The investigators will select two types of improved cookstoves to use in the feasibility trial.

The study design will be a crossover intervention trial in which all patients will first have a run-in observational period of 4 months with the traditional cookstove prior to randomization. At baseline, the investigators will obtain sociodemographic information for each household, respiratory outcomes and other health data for the participating women, and cooking times and practices including the types of fuels used. All 40 patients at each site will receive the two types of improved cookstoves, one after the other: 20 will be randomized to receive the first type of cookstove with a chimney and the other 20 to first receive the second type of improved cookstove with a chimney. The patients will be followed for 4 months before the crossover. The investigators will assess cooking behavioral practices and compliance with cookstove use monthly, and respiratory and environmental measures at the mid-point of the 4 month period to minimize carry-over effects. At the end of second 4 month period, the investigators will switch the order of the improved cookstoves and follow all participants for another 4 months. The investigators will assess behavior, compliance, respiratory and environmental measures as above. The study is expected to require 12 months to complete.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one woman aged 20 to 49 years who is the main cook.
* Have a traditional (i.e., open-fire) cookstove indoors with at least 3 walls and a roof.
* Are willing to have us install an improved cookstove and be willing to use it.
* Have household walls of mud, brick, cement, or wood.
* Capable of providing informed consent and responding to a questionnaire
* Full-time resident in the area

Exclusion Criteria:

* Have a new improved cookstove or a chimney in the household.
* Have household walls of thatch or bamboo no covered in mud.
* Plans to move from the area within one year.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Exposure to biomass fuel combustion | One year
  Measure change in levels of particulate matter concentrations and carbon monoxide between traditional cookstoves and improved, ventilated cookstoves in households in three rural populations in which biomass fuels are used almost exclusively for cooking.
Respiratory Outcomes | One year
  Measure change in respiratory outcomes (spirometry for FEV1 and peak expiratory flow, carboxyhemoglobin and DLCO) in women aged 20 to 49 years in three rural populations between traditional cookstoves and the improved, ventilated cookstoves.
Adoption process of improved cookstoves | One year
  Assess behaviors and attitudes in women 20-49 years of age in three rural populations regarding the adoption and continued use of improved cookstoves and evaluate the reasons for their preferred choice of cookstove at the end of the trial. Methodology includes: patient direct observations, in-depth interviews, semi-structured interviews and focus groups with study staff.

SECONDARY OUTCOMES:
Blood pressure | One year
  Measure change in blood pressure in women 20 to 49 years of age in three rural populations between traditional cookstoves and improved, ventilated cookstoves.

CONTACTS AND LOCATIONS:
Overall Officials: William Checkley, MD, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- Moi University, Eldoret, Kenya
- Nepal Nutrition Intervention Project - Sarlahi (NNIPS), Kathmandu, Nepal
- A.B. Prisma, Ayacucho, Ayacucho, Peru

REFERENCES:
- [Derived] Klasen E, Miranda JJ, Khatry S, Menya D, Gilman RH, Tielsch JM, Kennedy C, Dreibelbis R, Naithani N, Kimaiyo S, Chiang M, Carter EJ, Sherman CB, Breysse PN, Checkley W; COCINAS Trial Working Group. Feasibility intervention trial of two types of improved cookstoves in three resource-limited settings: study protocol for a randomized controlled trial. Trials. 2013 Oct 10;14:327. doi: 10.1186/1745-6215-14-327. PMID 24112419